CLINICAL TRIAL: NCT00215722
Title: XELOX Plus Cetuximab as First-Line Therapy in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo de Investigacao do Cancro Digestivo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GICR-P003
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

INTERVENTIONS:
Drug: Cetuximab

SUMMARY:
The first phase II trial with cetuximab and FOLFOX, as 1st line therapy for MCRC, presented at ASCO 2004, showed a 81% response rate, with no unexpected toxicities for the combination.

This study is aimed at establishing the efficacy and safety of the combination cetuximab/XELOX as first line therapy in patients with MCRC.

DETAILED DESCRIPTION:
The phase II trials with XELOX, demonstrated that is a highly effective first-line treatment for metastatic colorectal cancer, with response rates similar to the regimens with oxaliplatin and infusional 5-FU/LV (FOLFOX), but more convenient and likely to be preferred by both patients and health care providers.

Cetuximab has a significant anti-cancer activity in the setting of chemo-resistant disease which suggests that a much greater degree of benefit may ensue when it is used at an earlier stage of the disease course.

The first phase II trial with cetuximab and FOLFOX, as 1st line therapy for MCRC, presented at ASCO 2004, showed a 81% response rate, with no unexpected toxicities for the combination.

This study is aimed at establishing the efficacy and safety of the combination cetuximab/XELOX as first line therapy in patients with MCRC.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent, prior any study-specific procedures
* Male or female > = 18 years of age
* Histologically confirmed adenocarcinoma of the colon or rectum with metastatic disease not eligible for surgery with curative intent - in case of a unique metastatic lesion this should be confirmed by biopsy
* ECOG performance status < 1 at study entry
* Immunohistochemical evidence of EGFR expression on tumour tissue
* Presence of at least one unidimensional measurable lesion with a diameter > 20mm by conventional CT scan or MRI, and 10mm by spiral CT scan, according to the RECIST criteria (Index lesion(s) must not lie within an irradiated area)
* Have not received any Chemotherapy regimen for metastatic disease
* Life expectancy of > 3 months
* Neutrophils > = 1.5 x 109/L, platelet count > = 100 x 109/L, and haemoglobin > = 9 g/dL.
* Bilirubin level either normal or 1.5 x ULN
* ASAT and ALAT < = 2.5 x ULN (< = 5 x ULN in case of liver metastasis)
* Alkaline phosphatase < = 2.5 x ULN or < = 5 x ULN in case of liver metastasis or < = 10 x ULN in case of bone metastases
* Serum creatinine < = 1.5 x ULN or CrCl > 50 ml/min (Cockroft and Gault formula)
* Negative Pregnancy test within one week before treatment start, if applicable

Exclusion Criteria:

* Previous chemotherapy for metastatic CRC or adjuvant therapy with oxaliplatin or irinotecan.
* Adjuvant or neo-adjuvant therapy with 5 FU or derivatives is allowed if the chemotherapy treatment free interval is > 6 months and the patient have not progressed during treatment
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to study entry
* Prior radiotherapy is permitted if it was not administered to target lesions selected for this study
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to entry
* Previous exposure to EGFR-pathway targeting therapy
* History of evidence upon physical examination of CNS disease (e.g. primary brain tumour, seizure not controlled with standard therapy, any brain metastasis or history of stroke)
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease
* Pre-existing neuropathy > grade 1
* Known grade 3 or 4 allergic reaction to any of the components of the treatment.
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for > = 5 years will be allowed to enter the trial)
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Pregnant or lactating women
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome
* Known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Determine the Efficacy of the combination treatment (cetuximab plus capecitabine and oxaliplatin) as first-line therapy based on the overall response rate (ORR) according to the RECIST criteria.

SECONDARY OUTCOMES:
Determine the Safety parameters of combination treatment (cetuximab plus capecitabine and oxaliplatin) as first-line therapy analyzing the frequency, severity, duration and relationship of adverse events using the NCI CTCAE, version 3.0
Time to tumour progression (TTP)
Overall survival time (OS)
Evaluate the Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Evaristo Sanches, MD, Principal Investigator — Grupo de Investigação do Cancro Digestivo; Sérgio Barroso, MD, Principal Investigator — Grupo de Investigação do Cancro Digestivo
Locations (10):
- Portugal (10):
  - Hospital Garcia de Orta, Almada
  - Hospital Distrital do Barreiro, Barreiro
  - Hospital Distrital de Beja, Beja
  - Hospital de São Marcos, Braga
  - Hospitais da Universidade de Coimbra, Coimbra
  - IPO - Coimbra, Coimbra
  - Centro Hospitalar do Funchal, Funchal
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital do Divino Espírito Santo, Ponta Delgada
  - IPO - Porto, Porto